CLINICAL TRIAL: NCT05422950
Title: Relationship Between the Physical Condition and Functionality of Patients Post Intubation by Covid-19 With the Time of Stay in ICU an Stageof the Disease.
Brief Title: Relationship of Physical Condition and Functionality in Post-covid Patients
Status: Completed | Type: Observational
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Other Study IDs: 013-116
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: PHYSICAL ACTIVITY
Keywords: Covid-19; ICU; Physical deconditioning; Quality of life.
MeSH Terms: conditions — Motor Activity; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Relationship between physical condition and functionality in post-covid patients — Correlation study between the physical condition and functionality of patients after intubation due to covid 19

SUMMARY:
Cross-sectional, correlational cohort study where the variables Aerobic endurance (6-minute walk test), Muscle endurance (Medical research council MRC), Flexibility (Sit-and-reach test), Functionality (WHODAS 2.0), Number of days were analyzed hospitalized in the ICU, in post Covid-19 patients after one month of being discharged from the Intensive Care Unit. Users who met the criteria to be part of the research. For the analysis of variables and statistical significance of the results, the SPSS Statistics 22.0 program was used

DETAILED DESCRIPTION:
This research was developed in four phases:

Phase 1. Population selection The selection of post-intubated patients, who were discharged from the ICUs of Pasto in the months of June and July 2021, was made contact with patients and relatives two or three days before they are discharged from the ICU. One month after hospital discharge, the inclusion and non-inclusion criteria were contacted and verified, the study objectives were explained to patients and family members, then the informed consent was sent and completed. carried out the programming of the users for the respective data collection, the tests were carried out during the following month after being discharged from the ICU. The tests were carried out in person at the residence of each participant or that of the researcher. For the purposes of carrying out the tests, the patient had a companion in order to minimize the risks and ensure the correct application of the tests. Management and preparation guidelines for the tests were indicated to patients and family members.

Phase 2: Evaluation and data collection The population was assessed one month after being discharged. The researcher brought the necessary utensils to the agreed place for the execution of the tests. The study participants were verbally explained the objectives of the research, the procedure that was carried out and the signing of the informed consent was verified. Subsequently, the tests chosen by the researcher were evaluated and applied, taking into account aspects such as order, space and time.

Phase 3: Data tabulation and analysis Once the population data had been collected, the respective tabulation and analysis was carried out.

Phase 4: Results, discussion and conclusions Data analysis was performed to carry out the writing and analysis of the results, discussion, conclusions and limitations of the study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signature. Patients who have been in the ICU with a diagnosis of Covid-19. Post intubation patients due to Covid-19. Minimum 48 hours of stay in ICU. Maximum 2 months in ICU stay. Men and women between 18 and 60 years of age. Score according to Minmetal Test between 24 and 30. Patients who have undergone physical therapy during their hospitalization.

Exclusion Criteria:

* Cognitive impairment that does not allow order tracking. Patients with amputations. Present symptoms of SIRS. Being on supplemental oxygen. Those who die before the evaluation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study participants will be male and female patients of Colombian nationality, between the ages of 18 to 60 years post-intubated, who have been discharged between June and July 2021 in the intensive care units of the city of Pasto in the department of Nariño, diagnosed with Covid-19 by means of the C-reactive Protein test (CRP).
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
RELATIONSHIP BETWEEN THE PHYSICAL CONDITION AND FUNCTIONALITY OF PATIENTS POST INTUBATION BY COVID-19 WITH THE TIME OF STAY IN ICU AND STAGE OF THE DISEASE. | one year
  To evaluate the relationship between the days of stay in the ICU with the functionality and physical condition of the post-covid patients after hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Nacional, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No